CLINICAL TRIAL: NCT05260489
Title: Apollo Remote Observational Sleep Study
Status: Withdrawn | Type: Observational
Why Stopped: A similar dataset was being collected in another internal study.
Sponsor: Apollo Neuroscience, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AN001; 20214102 (Other: WCG IRB)
Record Dates: First submitted 2022-02-10; First posted 2022-03-02 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Sleep Quality; Heart Rate
Keywords: sleep quality, HRV, tvs, wearable
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to examine how Transcutaneous Vibratory Stimulation (TVS) produced by the Apollo wearable affects sleep and cardiovascular function in a diverse real-world population of Apollo users.

DETAILED DESCRIPTION:
The Apollo wearable is a consumer wellness device that offers a non-invasive, non-habit-forming wearable solution to improve performance and recovery under stress in children and adults by delivering gentle wave-like vibrations (Transcutaneous Vibratory Stimulation) to the body.

In this observational cohort study, we will assess sleep and cardiovascular metrics measured during sleep by Oura ring in participants who use Apollo wearable device both historically (2 years in the past) as well as in the future (two years forward). Participants will not be required to make any changes to their activities of daily living or lifestyle except for the continued use of their Apollo wearable devices and answer periodic questionnaires through an online survey tool.

Participant data for days with and without using the Apollo wearable will be analyzed to identify the near term and long term effects of using a TVS device on sleep and cardiovascular signatures. Environmental and confounding data will be derived from the survey data and biometrics data from the wearables.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or more
* Use both the Apollo wearable and Oura ring

Exclusion Criteria:

* Inability to complete questionnaires written in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Current Apollo Neuro customers who own and use Oura ring devices
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Average Heart Rate during sleep | Through study completion, an average of 4 years
  The average heart rate measured during sleep in beats per minute
Heart Rate Variability during sleep | Through study completion, an average of 4 years
  The Heart Rate Variability value measured during sleep in milli seconds
Lowest Heart Rate during sleep | Through study completion, an average of 4 years
  The lowest Heart Rate measured during sleep in beats per minutes
Sleep Onset | Through study completion, an average of 4 years
  The amount of time it takes to fall asleep once you are on the bed in seconds
Sleep efficiency | Through study completion, an average of 4 years
  The proportion of time spent sleeping to total time in bed
Wake time during sleep | Through study completion, an average of 4 years
  Total amount of time spent awake during a sleep session in seconds
Sleep duration | Through study completion, an average of 4 years
  Total amount of time spent sleeping in seconds
Deep sleep duration | Through study completion, an average of 4 years
  Total amount of time spent in deep sleep during sleep sessions in seconds
REM sleep duration | Through study completion, an average of 4 years
  Total amount of time spent in REM sleep during sleep sessions in seconds
Pittsburgh Sleep Quality Index (PSQI) | Through study completion, an average of 4 years
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. With a range of scores 1-21.

SECONDARY OUTCOMES:
Oura Sleep Score | Through study completion, an average of 4 years
  A proprietary Oura score (0-100) assigned to daily sleep based on sleep quality, age, gender, and sleep metrics.

CONTACTS AND LOCATIONS:
Overall Officials: David Rabin, MD PHD, Principal Investigator — Apollo Neuroscience, Inc.
Locations (1):
- Apollo Neuroscience, Inc., Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No